CLINICAL TRIAL: NCT03386162
Title: A Phase II Randomized Trial Comparing Alpelisib and Fulvestrant Versus Chemotherapy as Maintenance Therapy in Patients With PIK3CA Mutated Advanced Breast Cancer
Brief Title: SAFIR-PI3K A Phase II Randomized Maintenance Trial Comparing Alpelisib and Fulvestrant Versus Chemotherapy in PIK3CA Mutated Advanced Breast Cancer
Acronym: SAFIR-PI3K
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was halted Prematurely for low recruitment.
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0105/1701
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer, PI3K, Alpelisib
Keywords: Breast cancer, PI3K, alpelisib
MeSH Terms: conditions — Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — Alpelisib; Fulvestrant; Drug Therapy

STUDY DESIGN:
Intervention Model Description: In the randomized treatment phase, patients will be randomized 2:1 to receive:
  • Experimental arm (Arm A3): fulvestrant (500 mg intramuscular [as two 5 mL injections] every 28 days ± 3 days, with an additional injection on 15 after the first administration + Alpelisib (300 mg by mouth once daily, in a 21-day cycle). Premenopausal women will receive luteinizing hormone-releasing hormone (LH-RH) analogs in addition every 28 days ± 3 days.
  OR
  • Control arm (Arm B3): maintenance chemotherapy, meaning the same chemotherapy regimen used during the first 6-8 cycles (investigator's choice) or no antineoplastic treatment in case of toxicity after 4 full cycles.
  A total of approximately 90 patients will be enrolled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Arm A3) (Experimental): fulvestrant (500 mg intramuscular [as two 5 mL injections] every 28 days ± 3 days, with an additional injection on 15 after the first administration + Alpelisib (300 mg by mouth once daily, in a 21-day cycle). Premenopausal women will receive LH-RH analogs in addition every 28 days ± 3 days.
  Interventions: Drug: Alpelisib
- Control arm (Arm B3) (Active Comparator): maintenance chemotherapy, meaning the same chemotherapy regimen used during the first 6-8 cycles (investigator's choice) or no antineoplastic treatment in case of toxicity after 4 full cycles.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Alpelisib — fulvestrant (500 mg intramuscular [as two 5 mL injections] every 28 days ± 3 days, with an additional injection on 15 after the first administration + Alpelisib (300 mg by mouth once daily, in a 21-day cycle). Premenopausal women will receive LH-RH analogs in addition every 28 days ± 3 days.
  Other Names: fulvestrant
  Arms: Experimental arm (Arm A3)
Drug: Chemotherapy — maintenance chemotherapy, meaning the same chemotherapy regimen used during the first 6-8 cycles (investigator's choice) or no antineoplastic treatment in case of toxicity after 4 full cycles.
  Arms: Control arm (Arm B3)

SUMMARY:
SAFIR PI3K is an open-label multicenter phase II randomized trial, comparing alpelisib plus fulvestrant to maintenance chemotherapy in patient PIK3CA mutated with HR+/Her2- metastatic breast cancer who do not present progressive disease after 6-8 cycles of 1st or second line chemotherapy.

The primary objective is to determine whether treatment with alpelisib plus fulvestrant prolongs progression-free survival (PFS) compared to maintenance chemotherapy in patients PIK3CA mutated with hormone receptor positive (HR+), HER2-negative advanced breast cancer, who do not present a progressive disease after 6-8 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women (or men) with histologically confirmed metastatic breast cancer.
2. Hormone receptor positive (HR+) and no Her2 over-expression, according to local assessment.
3. Presence of PIK3CA mutation on exon 9 or 20, determined on metastatic tissue specimen (frozen or FFPE) or plasma (ctDNA). Eligible plasma should have been collected at time of metastatic disease progression and before to initiating chemotherapy.
4. Patient's disease is resistant to endocrine therapy (defined either as a relapse or progression occurred during endocrine therapy, whatever the line, or less than 12 months after the end of endocrine therapy in adjuvant context).
5. Patients who received 6 to 8 cycles of a first line chemotherapy, or patients who received 6 to 8 cycles of a first line stopped for progression followed by 6 to 8 cycles of a 2nd line chemotherapy, and who are presenting a stable or a responding disease at the time of randomization (4 full cycles of chemotherapy are accepted if stopped for toxicity reasons)
6. Age ≥18 years
7. WHO Performance Status 0/1
8. Presence of measurable or evaluable disease according to RECIST criteria v1.1
9. Patients will have had a wash-out period of at least 14 days for weekly (except monoclonal antibodies) or daily chemotherapies or 28 days for other chemotherapies from last chemotherapy administration prior to randomization and should have recovered from all residual toxicities (grade ≤1), excluding alopecia.
10. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

    1. Absolute Neutrophil Count (ANC) ≥1.5 x 10⁹/L
    2. Platelets ≥100 x 10⁹/L
    3. Hemoglobin ≥9.0 g/dL
    4. International normalized ratio (INR) ≤1.5
    5. Potassium, magnesium and calcium (corrected for albumin), within normal limits for the institution, or ≤Grade 1 severity according to NCI-CTCAE version 4.03 if judged clinically not significant by the investigator
    6. Serum creatinine ≤1.5 x upper limit of normal (ULN) or creatinine clearance ≥50 mL/min (Measured or calculated by Cockcroft and Gault formula)
    7. Total serum bilirubin ≤ ULN (or ≤1.5 x ULN if liver metastases are present; or total bilirubin ≤3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's Syndrome)
    8. Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤2.5 ULN (or <5.0 x ULN if liver metastases are present)
    9. Fasting plasma glucose (FPG) ≤140 mg/dL or ≤7.7 mmol/L* and Glycosylated Hemoglobin (HbA1c) ≤6.4% (both criteria have to be met).

       * For patients with FPG ≥100 mg/dL or HbA1c ≥5.7% (i.e. threshold for pre-diabetes) at baseline, recommend lifestyle changes according to ADA guidelines, i.e. dietary advice (e.g. small frequent meals, low carbohydrate content, high fiber, balancing carbohydrate intake over the course of the day, three small meals and 2 small snacks rather than one large meal) and exercise. A consultation with a diabetologist is highly recommended
11. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analysis
12. Patient with social insurance coverage.

Exclusion Criteria:

1. Spinal cord compression or symptomatic or progressive brain metastases (unless asymptomatic or treated and stable without steroids during the last 30 days).
2. Patient has received more than 2 previous lines of chemotherapy for metastatic disease before randomization.
3. Prior exposure to anthracyclines or mitoxantrone with cumulative exposure in excess of 360 mg/m² for doxorubicin, 720 mg/m² for epirubicin, or 72 mg/m² for mitoxantrone.
4. In the Investigator's judgment, patient has a life expectancy <3 months .
5. Disease progression occuring before randomization.
6. Patient has received prior treatment with any PI3K or AKT inhibitor (mTOR inhibitors are allowed)
7. Patient has history of hypersensitivity to any drugs or metabolites of similar chemical classes as alpelisib, or history of hypersensitivity to active or inactive excipients of any other study treatment.
8. Patient has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
9. Patient has received radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to randomization, and who has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia) or from whom ≥25% of the bone marrow was irradiated
10. Patient has participated to another clinical study with an investigational product during the last 30 days.
11. Patient has had major surgery within 14 days prior to starting study treatment or has not recovered from major side effects
12. Patient is currently receiving or has received systemic corticosteroids ≤2 weeks prior to starting study treatment, or has not fully recovered from side effects of such treatment
13. Patients with an established diagnosis of diabetes mellitus type I or not controlled type II, or documented steroid induced diabetes mellitus
14. Patient who necessitates to maintain the following drugs during study treatment :

    * Drugs known to be strong inhibitors or inducers of isoenzyme CYP3A4 including herbal medications (list of prohibited CYP3A4 inhibitors and inducers provided in Table 12)
    * Drugs with a known risk to induce Torsades de Pointes (list of prohibited QT prolonging drugs provided in Table 12) Note: The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the study treatment is initiated. Switching to a different medication prior to starting study treatment is allowed.
15. Patient is currently receiving warfarin or other coumarin derived anti-coagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed.
16. Patients who have other concurrent severe or uncontrolled medical conditions that would, in the Investigator's judgment, contraindicate patient participation in the individual patient program (eg. active or uncontrolled severe infection, chronic active hepatitis, immuno-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.)
17. Patient has currently documented pneumonitis
18. Patient has a known history of HIV infection (testing not mandatory)
19. Patient has any of the following cardiac abnormalities:

    * symptomatic congestive heart failure
    * history of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy
    * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
    * myocardial infarction ≤6 months prior to enrolment
    * unstable angina pectoris
    * serious uncontrolled cardiac arrhythmia
    * symptomatic pericarditis
    * QTcF >480 msec on the baseline ECG (using the QTcF formula) currently receiving treatment with medication that has a known risk to prolong the QT interval or inducing Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study treatment (list of prohibited QT prolonging drugs provided in Table 12)
20. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of any study treatment (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
21. Patient had previous or current malignancies of other histologies within the last 5 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin.
22. Pregnant or nursing (lactating) women.
23. Patient who does not accept to comply with highly effective contraception methods during the study treatment and through the duration as defined below after the final dose of study treatment:

    * Sexually active males should use a condom during intercourse while taking drug and for at least 4 weeks after the final dose of study treatment and should not father a child in this period.
    * Women of child-bearing potential must use highly effective contraception during study treatment and for at least 4 weeks after the final dose of study treatment and until resumption of menses (if longer than 4 weeks).
24. Patient has a history of non-compliance to medical regimen or inability to grant consent
25. Individuals deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 6 months
  To determine whether treatment with alpelisib plus fulvestrant prolongs progression-free survival (PFS) compared to maintenance chemotherapy in patients PIK3CA mutated with hormone receptor positive (HR+), HER2-negative advanced breast cancer, who do not present a progressive disease after 6-8 cycles of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Institut de Cancérologie de l'Ouest/Paul Papin, Angers
  - Institut Sainte-Catherine, Avignon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Chd Vendee, La Roche-sur-Yon
  - CHU Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CInstitut Regional du cancer-Centre Val D'Aurelle, Montpellier
  - Centre Eugène Marquis, Rennes
  - Centre Rene Huguenin, Saint-Cloud
  - Hôpitaux du Léman, Thonon-les-Bains
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif